CLINICAL TRIAL: NCT05969990
Title: Exploration of the Role of Tryptophan Metabolites in Pediatric Migraine
Brief Title: Tryptophan Metabolites in Pediatric Migraine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: QLCR20210182
Record Dates: First submitted 2023-05-15; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-01

CONDITIONS: Migraine in Children
Keywords: Migraine in Children, tryptophan metabolites

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: 100 children with migraine are included into case group and we will collect the blood of them to investigate tryptophan metabolites plasma concentration
  Interventions: Other: tryptophan metabolites in plasma
- control group: 100 healthy children are included into control group and we will collect the blood of them to investigate tryptophan metabolites plasma concentration
  Interventions: Other: tryptophan metabolites in plasma

INTERVENTIONS:
Other: tryptophan metabolites in plasma — we will investigate the tryptophan metabolites in plasma of children with migraine

SUMMARY:
Background:

Migraine is a common neurological disorder that also has a significant prevalence in children. Although the exact etiology of migraine is unknown, recent studies suggest an association between intestinal flora and migraine, and tryptophan metabolism is an important link between intestinal flora and the nervous system. However, the role of tryptophan metabolites in childhood migraine is not fully understood. Therefore, the aim of this study was to investigate the specific role of tryptophan metabolites in childhood migraine.

Study objectives:

The main objectives of this study were to assess the changes in tryptophan metabolites in childhood migraine and to explore their relationship with migraine attacks. Specific objectives include:

1. to determine the differences in tryptophan metabolites between children with migraine and healthy children;
2. to explore the correlation between tryptophan metabolites and migraine attacks
3. to assess the potential mechanisms of the role of tryptophan metabolites in childhood migraine.

Study methods:

1. participant recruitment: a certain number of pediatric migraine patients and healthy children were recruited as controls.
2. data collection: clinical information, medical history, and blood samples were collected from participants.
3. Tryptophan metabolite analysis: using appropriate experimental techniques, ELISA

Statistical analysis:

The main analyses included the following:

1. comparison of differences in tryptophan metabolites between migraine and control groups, using t-test or Wilcoxon rank sum test.
2. To assess the value of tryptophan metabolites in the diagnosis of migraine, ROC curve analysis was used to calculate the sensitivity, specificity, and AUC.
3. To explore the factors associated with tryptophan metabolites and migraine, multiple logistic regression analysis was used to assess the risk and protective effects of each factor on migraine.

Experimental hypothesis:

Our experimental hypothesis was that tryptophan metabolites may play a key role in the pathogenesis of childhood migraine, particularly kynurenine (KYN), quinolinic acid (QUINA), and kynurenic acid (KYNA). We hypothesized that in pediatric migraine patients, the concentrations of tryptophan metabolites would change significantly compared to healthy children. We further hypothesized that the concentrations of certain tryptophan metabolites correlate with the frequency and severity of migraine attacks. Based on these hypotheses, our study will examine tryptophan metabolite concentrations in blood samples and perform a comparative analysis between pediatric migraineurs and healthy children. We will also explore the correlation between tryptophan metabolites and migraine attacks and determine their risk and protective role in childhood migraine through multiple logistic regression analysis.

Outlook:

The results of this study are expected to reveal the important role of tryptophan metabolites in the pathogenesis of migraine in children and provide a new basis for the diagnosis and treatment of migraine in children. In addition, the study may also provide theoretical support for the development of relevant therapeutic strategies and interventions, and provide new ideas for the prevention and management of migraine in children.

DETAILED DESCRIPTION:
Method for determination of tryptophan metabolite content:

1. Timing of blood collection In the case group, blood was collected at any time during the first 2-4 hours of the migraine attack; in the inter-migraine attack group, blood was collected at least 24 hours before and after the headache-free period. In the healthy control group, blood was collected in a quiet state.
2. Storage and testing methods 5 ml of elbow venous blood was collected from patients and healthy children in purple tubes, and the samples were immediately transferred to ice-cold glass tubes containing a mixture of anticoagulant and protease inhibitor, and centrifuged at 3000 rpm for 5 minutes at 4°C. The supernatant was stored at -80°C, and tryptophan metabolite levels were measured by ELISA, and the case and control groups were compared and analyzed.

Feasibility analysis

1. The Elisa kit technology and medical statistics technology used in this project have been widely and maturely applied in other biomedical research fields, and the project has all the core technology reserves that can ensure the successful completion of the project.
2. The PICU of Qilu Hospital of Shandong University, which has rich experience in scientific research and clinical medicine, as well as rich clinical cases, is sufficient to meet the needs of scientific research; we have sufficient strength in terms of scientific research strength, talent demand and economic support to ensure the successful completion of our experiment.
3. The pediatric outpatient clinic of Qilu Hospital of Shandong University receives a large number of children with migraine every day, and the severity of the disease is complex and varied, so the number and diversity of children with migraine are sufficient to meet the needs of our experiment.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-18 years, male or female.
* Meet the ICHD-3 diagnostic criteria for migraine with aura, without aura, and chronic migraine.
* Migraine is diagnosed by two or more specialized neurologists.
* PedMIDAS score was more than 11.
* Migraine was never treated.
* Patients and family members gave informed consent to the study's purpose, significance, risks, benefits, and information of the study.

Exclusion Criteria:

* Presence of drug overdose.
* Autoimmune diseases.
* Neurological disorders other than migraine, intracranial masses.
* Congenital or genetic disorders.
* Diabetes, bronchial asthma, cardiovascular disease, pulmonary disease.
* Other types of primary and secondary headaches.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 100 children with migraine and 100 healthy children
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Tryptophan | In ictal period, during the first 2-4 hours of the attack. In interictal period, blood was collected at least 24 hours before and after the headache-free period. In the healthy group, blood was collected in the morning after fasting for eight hours.
Kynurenine | In ictal period, during the first 2-4 hours of the attack. In interictal period, blood was collected at least 24 hours before and after the headache-free period. In the healthy group, blood was collected in the morning after fasting for eight hours.
Kynurenic acid | In ictal period, during the first 2-4 hours of the attack. In interictal period, blood was collected at least 24 hours before and after the headache-free period. In the healthy group, blood was collected in the morning after fasting for eight hours.
Quinolinic acid | In ictal period, during the first 2-4 hours of the attack. In interictal period, blood was collected at least 24 hours before and after the headache-free period. In the healthy group, blood was collected in the morning after fasting for eight hours.
Serotonin | In ictal period, during the first 2-4 hours of the attack. In interictal period, blood was collected at least 24 hours before and after the headache-free period. In the healthy group, blood was collected in the morning after fasting for eight hours.

CONTACTS AND LOCATIONS:
Overall Officials: Xinjie Liu, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Junhui Liu, Jinan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kortesi T, Spekker E, Vecsei L. Exploring the Tryptophan Metabolic Pathways in Migraine-Related Mechanisms. Cells. 2022 Nov 27;11(23):3795. doi: 10.3390/cells11233795. PMID 36497053
- [Background] Curto M, Lionetto L, Negro A, Capi M, Perugino F, Fazio F, Giamberardino MA, Simmaco M, Nicoletti F, Martelletti P. Altered serum levels of kynurenine metabolites in patients affected by cluster headache. J Headache Pain. 2015;17(1):27. doi: 10.1186/s10194-016-0620-2. Epub 2016 Mar 22. PMID 27000870
- [Derived] Liu J, Xi K, Zhang L, Han M, Wang Q, Liu X. Tryptophan metabolites and gut microbiota play an important role in pediatric migraine diagnosis. J Headache Pain. 2024 Jan 5;25(1):2. doi: 10.1186/s10194-023-01708-9. PMID 38177986
- See also: Exploring the Tryptophan Metabolic Pathways in Migraine-Related Mechanisms — https://pubmed.ncbi.nlm.nih.gov/36497053/
- See also: Altered serum levels of kynurenine metabolites in patients affected by cluster headache. — https://pubmed.ncbi.nlm.nih.gov/27000870/

DOCUMENTS (2):
  • Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT05969990/SAP_000.pdf
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT05969990/ICF_001.pdf